CLINICAL TRIAL: NCT00360568
Title: Open-Label, 12-Month Safety and Efficacy Study of Levodopa - Carbidopa Intestinal Gel in Levodopa-Responsive Parkinson's Disease Subjects
Brief Title: Safety/Efficacy Study of Levodopa-Carbidopa Intestinal Gel in Parkinson's Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S187.3.003; 2006-000578-53 (EudraCT Number)
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Dyskinesias; Parkinson's Disease; Severe Motor Fluctuations
Keywords: carbidopa; severe motor fluctuations; intestinal gel; levodopa; efficacy; levodopa carbidopa intestinal gel; dyskinesia; Parkinson's Disease; Duodopa; levodopa-carbidopa; DUOPA
MeSH Terms: conditions — Dyskinesias; Parkinson Disease | interventions — Jejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Levodopa-Carbidopa Intestinal Gel (LCIG) (Experimental): All participants received LCIG, delivered through a percutaneous endoscopic gastrostomy with jejunal extension (PEG-J), administered for up to 12 months (52 weeks).
  Starting dose of LCIG was based on the participant's optimized oral levodopa-carbidopa dose that the subject was receiving just prior to randomization in Study S187.3.001 (NCT00357994) or Study S187.3.002 (NCT00660387), administered in the morning of the first day following Study Day 86 of either of these 2 previous studies. The LCIG infusion was expected to infuse over approximately16 hours each day with a rate of infusion within the range of 1 to 10 mL/hour (20 to 200 mg of levodopa/hour) in most instances.
  Interventions: Drug: Levodopa-carbidopa intestinal gel; Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: PEG tube; Device: J-tube

INTERVENTIONS:
Drug: Levodopa-carbidopa intestinal gel — Infusion should be kept within a range of 0.5-10 mL/hour (10-200 mg levodopa/hour) and is usually 2-6 mL/hour (40-120 mg levodopa/hour).
Device: CADD-Legacy® 1400 ambulatory infusion pump
Device: PEG tube — percutaneous endoscopic gastrostomy tube
Device: J-tube — jejunal tube

SUMMARY:
Long term safety and efficacy (12 months) of levodopa-carbidopa intestinal gel.

DETAILED DESCRIPTION:
Study S187.3.003 (NCT00360568) is a Phase 3, 12-month, open-label, multicenter continuation treatment study of the safety, tolerability, and efficacy of levodopa-carbidopa intestinal gel (LCIG) in the treatment of participants with levodopa-responsive Parkinson's disease (PD) with persistent motor fluctuations despite optimized treatment with available PD medications. All participants received LCIG.

Only participants who completed 12 weeks of double-blind, double-dummy treatment in Study S187.3.001 or S187.3.002 (NCT00357994/ NCT00660387) qualified for enrollment in this 12-month continuation treatment study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (PD) according to United Kingdon Parkinson's Disease Society (UKPDS) Brain Bank Criteria
* Levodopa-responsive with severe motor fluctuations
* Completion of protocol S187.3.001 (NCT00357994) or S187.3.002 (NCT00660387) and continue to meet the inclusion criteria for the preceding study

Exclusion Criteria:

* Patients with medically relevant abnormal findings (labs, electrocardiogram [ECG], physical examination, adverse events, psychiatric, neurological or behavioral disorders, etc.) at end of the double-blind phase (Week 12) of Study S187.3.001 (NCT00357994) or Study S187.3.002 (NCT00660387)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Benesh, Study Director — AbbVie
Locations (22):
- United States (16):
  - Site Reference ID/Investigator# 45869, Birmingham, Alabama
  - Site Reference ID/Investigator# 45834, Fountain Valley, California
  - Site Reference ID/Investigator# 45854, Los Angeles, California
  - Site Reference ID/Investigator# 45856, Oceanside, California
  - Site Reference ID/Investigator# 45859, Washington D.C., District of Columbia
  - Site Reference ID/Investigator# 45857, Bradenton, Florida
  - Site Reference ID/Investigator# 45863, Gainesville, Florida
  - Site Reference ID/Investigator# 45836, Port Charlotte, Florida
  - Site Reference ID/Investigator# 45874, Chicago, Illinois
  - Site Reference ID/Investigator# 45868, Lexington, Kentucky
  - Site Reference ID/Investigator# 45862, Baltimore, Maryland
  - Site Reference ID/Investigator# 45861, St Louis, Missouri
  - Site Reference ID/Investigator# 45873, New York, New York
  - Site Reference ID/Investigator# 45878, Cincinnati, Ohio
  - Site Reference ID/Investigator# 45850, Cleveland, Ohio
  - Site Reference ID/Investigator# 45887, Burlington, Vermont
- Germany (4):
  - Site Reference ID/Investigator# 45828, Bochum
  - Site Reference ID/Investigator# 45829, Bremerhaven
  - Site Reference ID/Investigator# 45825, Hanover
  - Site Reference ID/Investigator# 54402, Tübingen
- New Zealand (2):
  - Site Reference ID/Investigator# 45884, Auckland
  - Site Reference ID/Investigator# 45885, Hamilton

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- LCIG (Previous: LCIG + Placebo Capsules): All participants received levodopa-carbidopa intestinal gel (LCIG), delivered through a percutaneous endoscopic gastrostomy with jejunal extension (PEG-J), administered for up to 12 months (52 weeks). Starting dose of LCIG was based on the optimized oral levodopa-carbidopa dose that the participant was receiving just prior to randomization in Study S187.3.001 (NCT00357994) and Study S187.3.002 (NCT00660387), administered in the morning of the first day following Study Day 86 of these previous studies. The LCIG infusion was expected to infuse over approximately16 hours each day with a rate of infusion within the range of 1 to 10 mL/hour (20 to 200 mg of levodopa/hour) in most instances.
  In NCT00357994/NCT00660387 (previous study), these participants received double-blind, double-dummy treatment with LCIG + Placebo Capsules.
- LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules): All participants received LCIG, delivered through a PEG-J, administered for up to 12 months (52 weeks). Starting dose of LCIG was based on the optimized oral levodopa-carbidopa dose that the participant was receiving just prior to randomization in Study S187.3.001 (NCT00357994) and Study S187.3.002 (NCT00660387), administered in the morning of the first day following Study Day 86 of the previous studies. The LCIG infusion was expected to infuse over approximately16 hours each day with a rate of infusion within the range of 1 to 10 mL/hour (20 to 200 mg of levodopa/hour) in most instances.
  In NCT00357994/NCT00660387 (previous study), these participants received double-blind, double-dummy treatment with Placebo Gel + Levodopa-Carbidopa Capsules.
Period: Overall Study
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules)
Started | 33 | 29
Completed | 31 | 24
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- LCIG (Previous: LCIG + Placebo Capsules): All participants received LCIG, delivered through a PEG-J, administered for up to 12 months (52 weeks). Starting dose of LCIG was based on the optimized oral levodopa-carbidopa dose that the participant was receiving just prior to randomization in Study S187.3.001 (NCT00357994) and Study S187.3.002 (NCT00660387), administered in the morning of the first day following Study Day 86 of these previous studies. The LCIG infusion was expected to infuse over approximately16 hours each day with a rate of infusion within the range of 1 to 10 mL/hour (20 to 200 mg of levodopa/hour) in most instances.
  In NCT00357994/NCT00660387 (previous study), these participants received double-blind, double-dummy treatment with LCIG + Placebo Capsules.
- Total: Total of all reporting groups
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.0) | 64.8 (6.6) | 64.1 (7.9)
Age, Customized [Number; unit: participants]
  <65 years | 19 | 13 | 32
  >=65 years | 14 | 16 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths and Discontinuations Due to AEs
Description: AE=any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that: results in death; is life-threatening (an event in which the subject was at risk of death at the time of the event); requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or other important medical events. Treatment-emergent events (TEAE or TESAE)=those starting after the first dose of study drug. Severe=severity reported as 'severe' or missing. Possibly or Probably Treatment Related=drug-event relationship reported as 'possible', 'probable' or missing. Death=a fatal outcome of an SAE or AE.
Time Frame: From study enrollment to the end of study or early termination of treatment, including the removal of PEG-J, plus 30 days.
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion.
Measure: Number; unit: participants
Groups:
- LCIG (All Participants): All participants received LCIG, delivered through a PEG-J, administered for up to 12 months (52 weeks). Starting dose of LCIG was based on the optimized oral levodopa-carbidopa dose that the participant was receiving just prior to randomization in Study S187.3.001 (NCT00357994) and Study S187.3.002 (NCT00660387), administered in the morning of the first day following Study Day 86 of the previous studies. The LCIG infusion was expected to infuse over approximately 16 hours each day with a rate of infusion within the range of 1 to 10 mL/hour (20 to 200 mg of levodopa/hour) in most instances.
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants
  Deaths | 0 | 0 | 0
  TE Deaths | 0 | 0 | 0
  >=1 SAE | 5 | 9 | 14
  >=1 TESAE | 5 | 9 | 14
  >=1 TEAE Leading to Study Termination | 1 | 2 | 3
  >=1 TEAE | 31 | 28 | 59
  >=1 Severe TEAE | 5 | 10 | 15
  >=1 Possibly or ProbablyTreatment-Related TEAE | 28 | 20 | 48
  No TEAEs | 2 | 1 | 3

2. Primary Outcome: Number of Participants With Device Complications
Description: Complications of the infusion device were collected. Pump, intestinal tube, PEG, stoma, and other complications included (but were not limited to) device breakage, device leakage, device malfunction, device misuse, device occlusion, intentional and unintentional device removal by participant, complication of device insertion, device dislocation, device breakage, device dislocation, and device site reaction.
Time Frame: 12 months
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants
  >=1 Complication | 26 | 24 | 50
  Pump Complication | 18 | 16 | 34
  Intestinal Tube Complication | 15 | 16 | 31
  PEG Complication | 11 | 11 | 22
  Stoma Complication | 12 | 15 | 27
  Other | 6 | 4 | 10

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Values for Hematology Parameters
Description: Terms abbreviated in the table include females (f) and males (m).
Time Frame: 12 months
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion and had an assessment.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 28 | 61
participants
  Red Blood Cells <2.0 10^12/L (f); <2.5 10^12/L (m) | 0 | 0 | 0
  Haemoglobin <90 g/L (f); <100 g/L (m) | 0 | 1 | 1
  Haematocrit <30% (f); <34% (m) | 1 | 1 | 2
  White Blood Cells <2.8 10^9/L | 0 | 0 | 0
  White Blood Cells >16.0 10^9/L | 0 | 0 | 0
  Neutrophils, Absolute <1.2 10^9/L | 0 | 0 | 0
  Lymphocytes >80% | 0 | 0 | 0
  Lymphocytes, Absolute <.75 10^9/L | 2 | 0 | 2
  Eosinophils >10% | 0 | 0 | 0
  Monocytes >30% | 0 | 0 | 0
  Platelet Count <95 10^9/L | 0 | 0 | 0
  Platelet Count >700 10^9/L | 0 | 0 | 0
  Mean Corpuscular Volume <60 fL | 0 | 0 | 0
  Mean Corpuscular Volume >120 fL | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Values for Clinical Chemistry Parameters
Description: Terms abbreviated in the table include upper limit of normal (ULN), male (m), and female (f).
Time Frame: 12 months
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion; n=number of participants with an assessment.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants
  Sodium <126 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Sodium >156 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Albumin <25 g/L; n=27, 20, 47 | 0 | 0 | 0
  Albumin >70 g/L; n=27, 20, 47 | 0 | 0 | 0
  Potassium <3.0 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Potassium >6.0 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Creatinine >177 µmol/L; n=33, 28, 61 | 0 | 0 | 0
  Calcium <1.75 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Calcium >3.0 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Total Protein <45 g/L; n=33, 28, 61 | 0 | 0 | 0
  Total Bilirubin >2xULN; n=33, 28, 61 | 0 | 0 | 0
  Aspartate Aminotransferase >3xULN; n=33, 28, 61 | 0 | 0 | 0
  Alanine Aminotransferase >3xULN; n=33, 28, 61 | 0 | 0 | 0
  Gamma-glutamyl Transpeptidase >3x ULN;n=33, 28, 61 | 1 | 1 | 2
  Lactate dehydrogenase >3x ULN; n=33, 28, 61 | 0 | 0 | 0
  Alkaline Phosphatase >400 U/L; n=33, 28, 61 | 0 | 0 | 0
  Creatine Phosphokinase >3x ULN; n=33, 28, 61 | 0 | 0 | 0
  Non-fasting Glucose <2.78 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Non-fasting Glucose >16.0 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Uric Acid>500µmol/L(f);>590µmol/L(m);n=33, 28, 61 | 0 | 0 | 0
  Blood Urea Nitrogen >10.8 mmol/L; n=28, 22, 50 | 3 | 0 | 3
  Cholesterol >12.9 mmol/L; n=33, 28, 61 | 0 | 0 | 0
  Triglycerides >5.6 mmol/L; n=33, 28, 61 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Parameters
Description: Terms abbreviated in the table include supine systolic blood pressure (SuSBP), standing systolic blood pressure (StSBP), orthostatic systolic blood pressure (OSBP), supine diastolic blood pressure (SuDBP), standing diastolic blood pressure (StDBP), orthostatic diastolic blood pressure (ODBP), supine pulse (SuP) in beats per minute (bpm), standing pulse (StP), and body temperature (Temp). Increase and decrease are signified by ↑ and ↓, respectively.
Time Frame: 12 months
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion; n=number of participants with assessment.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants
  SuSBP <=90 and >30 mm Hg ↓ from BL; n=33, 29, 62 | 3 | 0 | 3
  SuSBP >=180 and >40 mm Hg ↑ from BL; n=33, 29, 62 | 1 | 2 | 3
  StSBP <=90 and >30 mm Hg ↓ from BL; n=33, 29, 62 | 4 | 7 | 11
  StSBP >=180 and >40 mm Hg ↑ from BL; n=33, 29, 62 | 0 | 0 | 0
  OSBP: ↓ >=30 mm Hg Supine to Standing; n=33,29,62 | 8 | 11 | 19
  SuDBP <=50 and >30 mm Hg ↓ from BL; n=33, 29, 62 | 0 | 1 | 1
  SuDBP >=105 and >30 mm Hg ↑ from BL; n=33, 29, 62 | 1 | 1 | 2
  StDBP <=50 and >30 mm Hg ↓ from BL; n=33, 29, 62 | 1 | 0 | 1
  StDBP >=105 and >30 mm Hg ↑ from BL; (n=33,29,62) | 2 | 1 | 3
  ODBP: ↓ >=20 mm Hg Supine to Standing; n=33,29,62 | 7 | 7 | 14
  SuP <=50 and >30 bpm ↓ from BL; n=33, 29, 62 | 1 | 0 | 1
  SuP >=120 and >30 bpm ↑ from BL; n=33, 29, 62 | 0 | 0 | 0
  StP <=50 and >30 bpm ↓ from BL; n=33, 29, 62 | 0 | 0 | 0
  StP >=120 and >30 bpm ↑ from BL; n=33, 29, 62 | 0 | 1 | 1
  Temp >=38.3° and >=1.1°C ↑ from BL; n=33, 29, 62 | 0 | 0 | 0
  Weight <=7% ↓ from BL; n=33, 27, 60 | 5 | 5 | 10
  Weight >=7% ↑ from BL; n=33, 27, 60 | 8 | 8 | 16

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Parameters
Description: Terms abbreviated in the table include heart rate (HR) in beats per minute (bpm), PR interval (PRI), QT interval corrected for heart rate using Bazett's formula (QTcB), and QT interval corrected for heart rate using Fridericia's formula (QTcF). Increase and decrease are signified by ↑ and ↓, respectively.
Time Frame: 12 months
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants
  HR <=50 and >30 bpm ↓ from BL; n=33, 28, 61 | 0 | 0 | 0
  HR >=120 and >30 bpm ↑ from BL; n=33, 28, 61 | 0 | 0 | 0
  PR Interval <120 msec; n=33, 27, 60 | 1 | 0 | 1
  PR Interval >220 msec; n=33, 27, 60 | 1 | 0 | 1
  QTcB Interval >480 msec; n=33, 27, 60 | 0 | 0 | 0
  QTcB Interval >60 msec ↑ from BL; n=33, 27, 60 | 0 | 0 | 0
  QTcF Interval >480 msec; n=33, 27, 60 | 0 | 0 | 0
  QTcF Interval >60 msec ↑ from BL; n=33, 27, 60 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Sleep Attacks at Baseline and Endpoint
Description: To prospectively monitor for the possible development of sleep attacks, participants were asked if they had experienced any events in which they fell asleep suddenly or unexpectedly, including while engaged in some activity (e.g., eating/drinking, speaking, or driving) or at rest, with or without any previous warning of sleepiness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants
  Participants with >=1 Sleep Attacks at Baseline | 0 | 0 | 0
  Participants with >=1 Sleep Attacks at Endpoint | 0 | 0 | 0

8. Primary Outcome: Summary of Minnesota Impulsive Disorder Interview (MIDI) Assessment of Intense Impulsive Behavior at Baseline (BL) and Post-baseline (PBL)
Description: The MIDI is a validated assessment of impulsive behavior consisting of a semistructured clinical interview assessing pathological gambling, trichotillomania (compulsive hair-pulling), kleptomania (compulsive stealing), pyromania (compulsive fire-setting), intermittent explosive disorder, compulsive buying, and compulsive sexual behavior.
Time Frame: Baseline, Post-baseline (up to Month 12)
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion; n=number of participants with assessment at timepoint.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants
  BL Pathological Gambling; n=33, 29, 62 | 0 | 0 | 0
  BL Trichotillomania; n=33, 29, 62 | 0 | 0 | 0
  BL Kleptomania; n=33, 29, 62 | 0 | 0 | 0
  BL Pyromania; n=33, 29, 62 | 0 | 0 | 0
  BL Intermittent Explosive Disorder; n=33, 29, 62 | 0 | 0 | 0
  BL Compulsive Buying; n=33, 29, 62 | 0 | 1 | 1
  BL Compulsive Sexual Behavior; n=33, 29, 62 | 0 | 1 | 1
  PBL Pathological Gambling; n=33, 27, 60 | 0 | 0 | 0
  PBL Trichotillomania; n=33, 27, 60 | 0 | 0 | 0
  PBL Kleptomania; n=33, 27, 60 | 0 | 0 | 0
  PBL Pyromania; n=33, 27, 60 | 0 | 0 | 0
  PBL Intermittent Explosive Disorder; n=33, 27, 60 | 0 | 0 | 0
  PBL Compulsive Buying; n=33, 27, 60 | 1 | 0 | 1
  PBL Compulsive Sexual Behavior; n=33, 27, 60 | 2 | 0 | 2

9. Primary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score at Endpoint
Description: The AIMS is an investigator-completed rating scale that has a total of 12 items rating involuntary movements of various areas of the participant's body. Items 1 through 10 are rated on a 5-point scale of severity from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), to 4 (severe), and items 11 and 12 are yes/no questions concerning problems with teeth or dentures. The total AIMS score was calculated by summing items 1-10, with a possible range of 0-40; a negative change indicates improvement. The AIMS was to be performed at consistent times, when the subject was experiencing his/her worst "On" time (dyskinesia [involuntary muscle movement]).
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
units on a scale
  Baseline; n=33, 29, 62 | 6.1 (6.0) | 5.3 (6.3) | 5.7 (6.1)
  Change from Baseline at Endpoint; n=33, 27, 60 | 6.1 (6.0) | 5.0 (6.3) | 5.6 (6.1)

10. Primary Outcome: Number of Participants With Confirmed Cases of Melanoma
Description: A comprehensive assessment for the presence of melanoma was performed during the screening period and at early termination/end of study by a dermatologist experienced with the diagnosis of the condition. If a suspicious lesion was present, a biopsy was obtained for proper diagnosis.
Time Frame: up to Month 12
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Clinically Significant Neurological Examination Findings
Description: The neurologic examination was to be done during "On" time. The neurological examination assessed: cranial nerves - assessment of cranial nerves II - XII, excluding fundoscopic examination; motor system - assessment of tone, strength, and abnormal movements; sensory system - including light touch, pinprick, joint position, and vibratory sense; reflexes - assessment of deep tendon reflexes and plantar responses (Babinski sign); coordination - assessment of upper and lower extremities; gait - assessment of base and tandem gait; station - assessment of posture and stability.
Time Frame: up to 12 months
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion and had a neurological examination.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 19 | 15 | 34
participants
  Cranial Nerve | 0 | 0 | 0
  Motor System | 3 | 2 | 5
  Sensory System | 2 | 1 | 3
  Reflexes | 1 | 1 | 2
  Coordination | 1 | 0 | 1
  Gait | 2 | 2 | 4
  Station | 2 | 2 | 4

12. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) Findings
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a systematically administered instrument developed to track suicidal adverse events across a treatment study. The instrument is designed to assess suicidal behavior and ideation, track and assess all suicidal events, as well as the lethality of attempts. Suicidal ideation categories include the following: wish to be dead; nonspecific active suicidal thoughts; active suicidal ideation without intent to act; active suicidal ideation with some intent to act but no plan; active suicidal ideation with plan and intent. Suicidal behavior categories include the following: actual attempt; interrupted attempt; aborted attempt; preparatory acts or behavior; suicidal behavior; completed suicide.
Time Frame: up to 12 months
Population: Safety Data Set: all enrolled participants who received at least one study S187-3-3003 LCIG infusion with a C-SSRS assessment during the study.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 12 | 7 | 19
participants
  Participants with Suicidal Ideations | 0 | 0 | 0
  Participants with Suicidal Ideations Only | 0 | 0 | 0
  Participants with Suicidal Behaviors | 0 | 0 | 0
  Participants with Suicidal Behaviors or Ideations | 0 | 0 | 0

13. Primary Outcome: Number of Participants Taking at Least 1 Concomitant Medication During the Study
Description: Concomitant medications include medications started on or after the first open-label LCIG infusion as well as medications started prior to the first open-label infusion but continued during the study.
Time Frame: 12 months
Population: Safety Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion.
Measure: Number; unit: participants
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
participants | 33 | 29 | 62

14. Secondary Outcome: Change From Baseline in Average Daily "Off" Time at Endpoint
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. Negative change from baseline for "off" time indicates improvement.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: Full Analysis Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion and had data for baseline and at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 32 | 27 | 59
hours
  Baseline | 2.87 (2.18) | 5.18 (2.05) | 3.92 (2.40)
  Change from Baseline at Endpoint | -0.42 (2.67) | -2.34 (2.78) | -1.30 (2.86)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

15. Secondary Outcome: Change From Baseline in Average Daily Normalized "On" Time With Troublesome Dyskinesia at Endpoint
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 32 | 27 | 59
hours
  Baseline | 1.09 (2.07) | 0.82 (1.54) | 0.97 (1.84)
  Change from Baseline at Endpoint | -0.58 (2.18) | 0.15 (2.17) | -0.24 (2.19)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.394, t-test, 2 sided

16. Secondary Outcome: Change From Baseline in Average Daily "On" Time Without Troublesome Dyskinesia at Month 12
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. "On" time without troublesome dyskinesia (involuntary muscle movement) is defined as "on" time without dyskinesia and "on" time with non-troublesome dyskinesia. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. Positive change from Baseline for "on" time without troublesome dyskinesia indicates improvement.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 32 | 27 | 59
hours
  Baseline | 12.04 (2.42) | 10.00 (2.62) | 11.11 (2.69)
  Change from Baseline at Endpoint | 1.00 (2.58) | 2.19 (3.70) | 1.54 (3.17)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

17. Secondary Outcome: Clinical Global Impression - Status (CGI-S) Score at Baseline and Clinical Global Impression - Improvement (CGI-I) Score at Endpoint
Description: The CGI-S is a global assessment by the Investigator of current symptomatology and impact of illness on functioning. The ratings of the CGI-S are as follows: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, and 7 = among the most extremely ill. The CGI-I is a global assessment by the Investigator of the change in clinical status since the start of treatment. The CGI-I ratings are as follows: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: Full Analysis Data Set: all enrolled participants who received at least one study S187.3.003 LCIG infusion and had data for baseline and at least 1 post-baseline assessment; n=number of participants with assessment at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 29 | 62
units on a scale
  CGI-S at Baseline; n=32, 28, 60 | 3.0 (1.3) | 3.7 (1.3) | 3.3 (1.3)
  CGI-I at Endpoint; n=33, 29, 62 | 2.1 (1.2) | 2.3 (1.6) | 2.2 (1.4)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

18. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part I Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part I Score is the sum of the answers to the 4 questions that comprise Part I, each of which are measured on a 5-point scale (0-4). The Part I score ranges from 0-16 and higher scores are associated with more disability.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 1.6 (1.8) | 1.2 (1.0) | 1.4 (1.5)
  Change from Baseline at Endpoint | 0.3 (1.9) | 0.7 (1.7) | 0.5 (1.8)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.055, t-test, 2 sided

19. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to the 13 questions that comprise Part II, each of which are measured on a 5-point scale (0-4). The Part II score ranges from 0-52 and higher scores are associated with more disability.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 8.6 (6.5) | 12.1 (7.0) | 10.1 (6.9)
  Change from Baseline at Endpoint | 0.5 (3.4) | -1.0 (7.0) | -0.2 (5.3)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.766, t-test, 2 sided

20. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part III score is the sum of the 27 answers provided to the 14 Part III questions, each of which are measured on a 5-point scale (0-4). The Part III score ranges from 0-108 and higher scores are associated with more disability.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 25 | 58
units on a scale
  Baseline | 16.2 (12.7) | 19.0 (10.5) | 17.4 (11.8)
  Change from Baseline at Endpoint | 1.5 (7.0) | -0.5 (10.4) | 0.6 (8.6)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.571, t-test, 2 sided

21. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Total Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The total score is the sum of the responses to the 31 questions (44 answers) that comprise Parts I-III of the scale. The total score will range from 0-176, with 176 representing the worst (total) disability, and 0 representing no disability.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 25 | 58
units on a scale
  Baseline | 26.4 (18.9) | 32.4 (16.1) | 29.0 (17.8)
  Change from Baseline at Endpoint | 2.3 (9.0) | -1.0 (15.0) | 0.9 (12.0)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.583, t-test, 2 sided

22. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part IV Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part IV Score is the sum of the answers to the 11 questions that comprise Part IV, each of which are measured on a 5-point scale (0-4) or a 2-point scale (0 or 1). The Part IV score ranges from 0-23 and higher scores are associated with more disability.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 5.8 (2.7) | 7.0 (3.2) | 6.3 (3.0)
  Change from Baseline at Endpoint | -1.6 (2.5) | -1.4 (3.0) | -1.5 (2.7)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

23. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Summary Index at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. These include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The PDQ-39 Summary Index is the sum of all answers divided by the highest score possible (i.e. number of answers multiplied by 4) which is multiplied by 100 to put the score on a 0-100 scale. Higher scores are associated with more severe symptoms.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 32 | 26 | 58
units on a scale
  Baseline | 22.2 (17.3) | 32.8 (17.0) | 26.9 (17.8)
  Change from Baseline at Endpoint | 1.5 (12.7) | -3.5 (13.4) | -0.7 (13.2)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.670, t-test, 2 sided

24. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Mobility Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Mobility (e.g., fear of falling when walking) includes 10 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 27.6 (24.1) | 43.8 (25.4) | 34.7 (25.8)
  Change from Baseline at Endpoint | 2.3 (19.5) | -8.5 (18.6) | -2.5 (19.7)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.341, t-test, 2 sided

25. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Activities of Daily Living Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Activities of Daily Living (e.g., difficulty cutting food) includes 6 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 25.9 (24.8) | 39.4 (21.3) | 31.9 (24.1)
  Change from Baseline at Endpoint | 0.4 (14.0) | -6.7 (19.9) | -2.8 (17.1)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.220, t-test, 2 sided

26. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Emotional Well-Being Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Emotional Well-being (e.g., feelings of isolation) includes 6 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 32 | 26 | 58
units on a scale
  Baseline | 20.1 (20.3) | 26.3 (17.2) | 22.8 (19.1)
  Change from Baseline at Endpoint | 4.0 (16.4) | 1.9 (18.1) | 3.1 (17.1)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.174, t-test, 2 sided

27. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Stigma Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Stigma (e.g., social embarrassment) consists of 4 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 32 | 26 | 58
units on a scale
  Baseline | 16.4 (21.3) | 23.8 (19.0) | 19.7 (20.5)
  Change from Baseline at Endpoint | 0.2 (15.2) | -6.3 (20.7) | -2.7 (18.0)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.259, t-test, 2 sided

28. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Social Support Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Social Support includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 11.9 (18.2) | 17.1 (17.8) | 14.2 (18.0)
  Change from Baseline at Endpoint | 1.8 (17.2) | -2.7 (15.5) | -0.2 (16.5)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.922, t-test, 2 sided

29. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Cognition Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Cognition includes 4 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 15.0 (14.1) | 24.8 (18.9) | 19.3 (16.9)
  Change from Baseline at Endpoint | 1.3 (16.3) | 3.8 (16.7) | 2.4 (16.4)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.258, t-test, 2 sided

30. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Communication Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Communication includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 15.9 (16.3) | 31.7 (23.2) | 22.9 (21.0)
  Change from Baseline at Endpoint | 8.3 (18.4) | -1.9 (15.3) | 3.8 (17.7)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.104, t-test, 2 sided

31. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Bodily Discomfort Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Bodily Discomfort includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Endpoint | 32.1 (25.8) | 34.9 (22.9) | 33.3 (24.4)
  Change from Baseline at Endpoint | -2.8 (18.8) | 1.0 (19.5) | -1.1 (19.0)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.650, t-test, 2 sided

32. Secondary Outcome: Change From Baseline in EuroQol Quality of Life Scale (EQ-5D) Summary Index at Endpoint
Description: The EQ-5D is a participant answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that essentially attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 to 1.00 with positive change indicating improvement.
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 0.778 (0.144) | 0.676 (0.158) | 0.733 (0.158)
  Change from Baseline at Endpoint | -0.009 (0.173) | -0.006 (0.220) | -0.008 (0.193)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.759, t-test, 2 sided

33. Secondary Outcome: Change From Baseline in EuroQol Quality of Life Scale (EQ-5D) Visual Analogue Scale (VAS) at Endpoint
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where 100 is the 'best imaginable health state' and 0 is the 'worst imaginable health state.'
Time Frame: Baseline, Endpoint (Month 12 or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 33 | 26 | 59
units on a scale
  Baseline | 76.7 (16.2) | 62.1 (22.0) | 70.2 (20.2)
  Change from Baseline at Endpoint | -0.9 (15.1) | 4.5 (15.5) | 1.5 (15.4)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.459, t-test, 2 sided

34. Secondary Outcome: Change From Baseline in Zarit Burden Interview (ZBI) Total Score at Endpoint
Description: The ZBI is a 22-item questionnaire regarding the caregiver/subject relationship and evaluates the caregiver's health condition, psychological well-being, finances and social life. Each question is answered on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=quite frequently, and 4=nearly always). The caregiver burden is evaluated by the total score (range 0 to 88) obtained from the sum of the answers to the 22 questions. Higher scores are associated with a higher level of burden for the caregiver.
Time Frame: Baseline, Endpoint (Month 12 months or last post-baseline visit)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Number analyzed (Participants) | 24 | 20 | 44
units on a scale
  Baseline | 22.1 (15.3) | 27.0 (17.2) | 24.3 (16.2)
  Change from Baseline at Endpoint | 1.1 (9.7) | -1.8 (9.0) | -0.2 (9.4)
Statistical Analysis 1: Comparison: LCIG (All Participants); Test type: Superiority or Other; p = 0.899, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From study enrollment to the end of study or early termination of treatment, including the removal of PEG-J (up to 52 weeks), plus 30 days.
Description: Serious AEs and treatment-emergent AEs are presented. Treatment-emergent AEs were defined as AEs that began or worsened from date of the first dose of study drug in this study to the end of therapy (last dose of study drug or PEG-J removal, whichever is later) plus 30 days.
Arm/Group | LCIG (Previous: LCIG + Placebo Capsules) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) | LCIG (All Participants)
Serious Adverse Events (participants affected / at risk) | 5/33 | 9/29 | 14/62
Other Adverse Events (participants affected / at risk) | 29/33 | 26/29 | 55/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCIG (Previous: LCIG + Placebo Capsules) (N=33) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) (N=29) | LCIG (All Participants) (N=62)
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 2
FAECALOMA (Gastrointestinal disorders) | 0 | 1 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 1 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 1
PERITONITIS (Gastrointestinal disorders) | 0 | 1 | 1
ASTHENIA (General disorders) | 1 | 1 | 2
COMPLICATION OF DEVICE INSERTION (General disorders) | 1 | 2 | 3
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 1
PNEUMONIA (Infections and infestations) | 0 | 2 | 2
SEPSIS (Infections and infestations) | 0 | 1 | 1
GASTROINTESTINAL INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 1
COLONOSCOPY (Investigations) | 0 | 1 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 1
DELUSION (Psychiatric disorders) | 0 | 1 | 1
HALLUCINATION (Psychiatric disorders) | 0 | 1 | 1
HALLUCINATION, AUDITORY (Psychiatric disorders) | 0 | 1 | 1
PARANOIA (Psychiatric disorders) | 0 | 1 | 1
RENAL MASS (Renal and urinary disorders) | 0 | 1 | 1
URETHRAL STENOSIS (Renal and urinary disorders) | 1 | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCIG (Previous: LCIG + Placebo Capsules) (N=33) | LCIG (Previous: Placebo Gel + Levodopa-Carbidopa Capsules) (N=29) | LCIG (All Participants) (N=62)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 0 | 3
CONSTIPATION (Gastrointestinal disorders) | 4 | 5 | 9
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 4
NAUSEA (Gastrointestinal disorders) | 4 | 5 | 9
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 | 2 | 2
VOMITING (Gastrointestinal disorders) | 2 | 3 | 5
COMPLICATION OF DEVICE INSERTION (General disorders) | 2 | 0 | 2
FATIGUE (General disorders) | 0 | 2 | 2
OEDEMA PERIPHERAL (General disorders) | 2 | 1 | 3
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 5 | 6 | 11
RHINITIS (Infections and infestations) | 0 | 2 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 0 | 3
URINARY TRACT INFECTION (Infections and infestations) | 5 | 4 | 9
CONTUSION (Injury, poisoning and procedural complications) | 4 | 1 | 5
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 2 | 2
FALL (Injury, poisoning and procedural complications) | 7 | 6 | 13
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 | 2 | 2
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 7 | 11 | 18
LACERATION (Injury, poisoning and procedural complications) | 1 | 2 | 3
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 3 | 5 | 8
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 2 | 3
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 4 | 3 | 7
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 2 | 3 | 5
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 | 2 | 3
BLOOD HOMOCYSTEINE INCREASED (Investigations) | 5 | 2 | 7
VITAMIN B6 DECREASED (Investigations) | 8 | 5 | 13
WEIGHT DECREASED (Investigations) | 2 | 3 | 5
X-RAY ABNORMAL (Investigations) | 2 | 0 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 2 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 2 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 8
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 2 | 0 | 2
DISTURBANCE IN ATTENTION (Nervous system disorders) | 2 | 0 | 2
DYSKINESIA (Nervous system disorders) | 4 | 3 | 7
DYSTONIA (Nervous system disorders) | 1 | 4 | 5
FREEZING PHENOMENON (Nervous system disorders) | 4 | 3 | 7
HEADACHE (Nervous system disorders) | 5 | 1 | 6
PARKINSON'S DISEASE (Nervous system disorders) | 4 | 4 | 8
POLYNEUROPATHY (Nervous system disorders) | 3 | 3 | 6
RESTLESS LEGS SYNDROME (Nervous system disorders) | 2 | 2 | 4
ABNORMAL DREAMS (Psychiatric disorders) | 0 | 2 | 2
ANXIETY (Psychiatric disorders) | 3 | 2 | 5
DEPRESSION (Psychiatric disorders) | 3 | 2 | 5
HALLUCINATION (Psychiatric disorders) | 1 | 2 | 3
INSOMNIA (Psychiatric disorders) | 2 | 7 | 9
SLEEP ATTACKS (Psychiatric disorders) | 0 | 3 | 3
POLLAKIURIA (Renal and urinary disorders) | 3 | 0 | 3
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 2 | 4 | 6
LENTIGO (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
RASH (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 3 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.